CLINICAL TRIAL: NCT06352892
Title: A Phase 1, Open-label, Randomized, Parallel-group, Single-dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of AMG 133 Administered Subcutaneously in Chinese Subjects With Obesity or Overweight
Brief Title: A Study to Evaluate AMG 133 in Chinese Participants With Obesity or Overweight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210201
Record Dates: First submitted 2024-04-03; First posted 2024-04-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Obesity
Keywords: Obesity; Overweight; AMG 133
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Maridebart Cafraglutide Dose 1 (Experimental): Participants will receive a single SC lower dose of Maridebart Cafraglutide.
  Interventions: Drug: Maridebart Cafraglutide
- Group 2: Maridebart Cafraglutide Dose 2 (Experimental): Participants will receive a single SC higher dose of Maridebart Cafraglutide.
  Interventions: Drug: Maridebart Cafraglutide

INTERVENTIONS:
Drug: Maridebart Cafraglutide — Solution for SC injection.
  Other Names: AMG 133

SUMMARY:
The main objective of the study is to assess the pharmacokinetics (PK) of Maridebart Cafraglutide after a single subcutaneous (SC) administration in overweight or obese Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed informed consent.
* Participants must be of Chinese ancestry with biological parents and all 4 grandparents of Chinese ancestry.
* Male or female participants, between 18 and 65 years of age (inclusive) at the time of Screening. Female participants must be of nonchildbearing potential.
* Except for obesity, no clinically significant findings from medical history (that requires the use of medications and/or treatment), physical examination, 12-lead electrocardiogram (ECG), vital signs measurements, and clinical laboratory evaluations.
* Body mass index between 24 and 40 kg/m^2 (inclusive) at the time of Screening.
* Have a stable body weight (<5 kg self-reported change) within 3 months before Screening.
* Have not modified diet or adopted any nutritional lifestyle modification for 3 months.

Exclusion Criteria:

* History or evidence, at Screening or Check-in, of clinically significant disorder, condition, or disease not otherwise excluded that, in the opinion of the Investigator (or designee), would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.
* History or evidence, at Screening, of diabetes (regardless of type), based on Hemoglobin A1C of > 7%.
* History or evidence of endocrine disorder (such as Cushing's Syndrome) that can cause obesity.
* Previous surgical procedure for obesity (excluding liposuction if performed >1 year before study entry) within past 6 months from Check-in.
* History or current signs or symptoms of cardiovascular disease.
* History of clinically significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee) and in consultation with the Sponsor.
* Estimated glomerular filtration rate less than at least 60 mL/min/1.73 m^2 at Screening or Check-in.
* Alanine aminotransferase or aspartate aminotransferase >2 x the upper limit of normal at Screening or Check-in.
* Positive hepatitis B or hepatitis C panel and/or positive human immunodeficiency virus test at Screening. Participants whose results are compatible with prior immunity (vaccination or prior infection) may be included.
* Use of any over-the-counter or prescription medications within 30 days or 5 half-lives (whichever is longer) before Check-in.

  1. Acetaminophen (paracetamol; up to 2 g per day) for analgesia will be allowed.
  2. Hormone replacement therapy (eg, estrogen, thyroid) will be allowed.
* Current or prior use of any glucagon-like peptide 1 agonist within the past 3 months prior to Check-in.
* All herbal medicines (eg, St. John's wort), Traditional Chinese Medicine herbs or formulations, vitamins, and supplements consumed by the participant within the 30 days prior to enrollment, unless deemed acceptable by the Investigator (or designee) and in consultation with the Sponsor.
* History of alcoholism or regular alcohol consumption of >14 units per week for males and >7 units for females or drug/chemical abuse within 1 year prior to Check-in.
* Alcohol consumption from 48 hours prior to Check-in and is unwilling to limit alcohol intake to a maximum of 1 unit/day on all other days, while not in the clinical research unit, from Screening through the End of Study (EOS) visit.
* Use of tobacco- or nicotine-containing products within 6 months prior to Check-in.
* Female participants with a positive pregnancy test at Screening or Check-in.
* Female participants lactating/breastfeeding or who plans to breastfeed during the study through 90 days after the EOS visit.
* Unwilling to adhere to contraceptive requirements through 90 days after the EOS visit.
* Male participants with a female partner of childbearing potential and not willing to inform his partner of his participation in this clinical study.
* Pregnant partner (of a male participant) or partner planning to become pregnant who is unwilling to practice abstinence (refrain from heterosexual intercourse) or use contraception while the participant is on study through 90 days after the EOS visit.
* Participant has received a dose of an investigational drug within the past 90 days or 5 half-lives, whichever is longer, prior to Check-in.
* Have previously completed or withdrawn from this study or any other study investigating Maridebart Cafraglutide or have previously received the investigational product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Maridebart Cafraglutide | Up to approximately 120 days
Area Under the Plasma Concentration-time Curve (AUC) from Time Zero to the Last Quantifiable Concentration (AUClast) of Maridebart Cafraglutide | Up to approximately 120 days
AUC from Time Zero Extrapolated to Infinity (AUCinf) of Maridebart Cafraglutide | Up to approximately 120 days

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events | Up to approximately 120 days
Number of Participants with Serious Adverse Events | Up to approximately 120 days
Number of Participants with Anti-Maridebart Cafraglutide Antibodies | Up to approximately 120 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com